CLINICAL TRIAL: NCT03284411
Title: Spinal Cord Stimulation (SCS) Dosing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17046
Record Dates: First submitted 2017-08-31; First posted 2017-09-15 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Back Pain; Leg Pain
MeSH Terms: conditions — Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spinal Cord Stimulation (Experimental): Each subject was programmed to 4 different amplitude settings: 80%, 60%, 40% and 20% of perception threshold amplitude
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Programming

SUMMARY:
This study characterized the effects of amplitude on subject satisfaction and pain relief in subjects being treated by SCS.

DETAILED DESCRIPTION:
This feasibility study assessed the following outcomes:

* Patient satisfaction
* VAS pain scores

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older
2. Implanted with a RestoreSensor system (for back and leg pain) for at least 1 month
3. Has approproate SCS settings
4. Willing and able to provide signed and dated informed consent
5. Capable of comprehending and consenting in English
6. Capable of getting into the supine and sitting positions
7. Willing and able to comply with all study procedures and visits
8. On stable (no change in dose, route, or frequency) prescribed pain medications

Exclusion Criteria:

1. Implanted with leads for peripheral nerve stimulation or an implantable intrathecal drug delivery system
2. Had a pain-related surgery in the previous 1 month of enrollment or the intent to undergo surgery during the period of the study
3. Implanted with quadripolar lead
4. Currently enrolled or planning to enroll in a potentially confounding clinical study during the course of the study
5. Pregnant or is of child-bearing potential and unwilling to use a medically acceptable form of birth control during the study
6. Has untreated major psychiatric comorbidity
7. Has serious drug-related behavioral issues
8. Has unresolved major issues of secondary gain

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Arizona Pain Doctors, Chandler, Arizona
  - Georgia Pain and Wellness Center, Lawrenceville, Georgia
  - Global Scientific Innovations, Evansville, Indiana
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Kentuckiana Pain Specialists, Louisville, Kentucky
  - Drez One, LLC, Somerset, Kentucky
  - Regional Brain & Spine, Cape Girardeau, Missouri
  - Precision Spine Care, Tyler, Texas
  - Northwest Pain Care, Inc., Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation: Each subject was programmed to 4 different amplitude settings (80, 60, 40, and 20 percent of their perception threshold amplitude).
  Spinal Cord Stimulation: Programming
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Spinal Cord Stimulation: Each subject was programmed to 4 different amplitude settings (80, 60, 40, and 20 percent of their perception threshold).
  Spinal Cord Stimulation: Programming
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: SCS Therapy Satisfaction
Description: To characterize the effect of four different amplitude settings on baseline SCS therapy satisfaction. At each follow-up visit, the following question was asked to measure satisfaction: "Overall how satisfied or unsatisfied are you with this therapy?". The response choices were as follows: "very satisfied", "somewhat satisfied", "neutral", "somewhat unsatisfied", "very unsatisfied". Each subject was considered to have maintained their baseline SCS therapy satisfaction if they selected the response "very satisfied", "somewhat satisfied", or "neutral", otherwise they were considered dissatisfied with the therapy. The first visit in which each subject reported dissatisfaction of the therapy was recorded. The amplitude used during the prior visit was then considered to be the minimum amplitude that maintained each subject's therapy satisfaction. The frequency and percentage of subjects' that maintained baseline satisfaction were reported at each amplitude level.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Spinal Cord Stimulation: Each subject was programmed to 4 different amplitude settings (80, 60, 40, and 20 percent of perception threshold).
  Spinal Cord Stimulation: Programming
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 30
Participants
  Baseline | 6
  80% perception threshold | 2
  60% perception threshold | 1
  40% perception threshold | 0
  20% perception threshold | 21

2. Secondary Outcome: Number of Participants Maintaining Baseline Pain as Measured on the Visual Analog Scale (VAS)
Description: To characterize the effect of four different amplitude settings on baseline pain relief. During each follow-up period the VAS pain score was recorded once a day, on a multi-day diary, where subjects rated their pain by making a vertical slash mark through the 0-10 cm line that best described their pain during the last 24 hours, with 0 = No pain and 10 = Worst pain imaginable. The higher VAS pain score represented worse pain. The average VAS pain scores from the last 3 days of the diary prior to the scheduled visit was used for analysis. Each subject was considered to have maintained their baseline pain if there was less than a 2 point increase in their average pain score at the follow-up period. The amplitude used during the prior visit was then considered to be the minimum amplitude that maintained the subject's pain relief. The frequency and percentage of subjects' that maintained their average baseline VAS pain score were reported at each amplitude level.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Spinal Cord Stimulation: Each subject was programmed to 4 different amplitude settings (80, 60, 40, 20 percent of perception threshold).
  Spinal Cord Stimulation: Programming
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 30
Participants
  Baseline | 5
  80% perception threshold | 3
  60% perception threshold | 1
  40% perception threshold | 2
  20% perception threshold | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study discontinuation with an average of 2.2 months
Groups:
- Spinal Cord Stimulation: Each subject was programmed to 4 different amplitude settings (80, 60, 40, and 20 percent of their perception threshold)
  Spinal Cord Stimulation: Programming
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (N=30)
Device stimulation issue (Product Issues) | 3 (3)
Inadequate analgesia (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03284411/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03284411/SAP_001.pdf